CLINICAL TRIAL: NCT04875416
Title: Phenotype, Genotype and Biomarkers 2
Acronym: PGB2
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Michael Benatar, Professor, University of Miami
Other Study IDs: 20200888; U54NS092091 (NIH)
Record Dates: First submitted 2021-04-14; First posted 2021-05-06 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis; Hereditary Spastic Paraplegia; Primary Lateral Sclerosis; Progressive Muscular Atrophy; Frontotemporal Dementia
Keywords: ALS; PLS; PMA; HSP; FTD; MSP
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Spastic Paraplegia, Hereditary; Motor Neuron Disease; Muscular Atrophy, Spinal; Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine and CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary participants: Patients that have or are suspected to have ALS or a related neurodegenerative disease
- Secondary Participants: Family members of primary participants enrolled in the study

SUMMARY:
The purpose of this study is to learn more about amyotrophic lateral sclerosis (ALS) and other related neurodegenerative diseases, including frontotemporal dementia (FTD), primary lateral sclerosis (PLS), hereditary spastic paraplegia (HSP), progressive muscular atrophy (PMA) and multisystem proteinopathy (MSP). More precisely, the investigator wants to identify the links that exist between the disease phenotype (phenotype refers to observable signs and symptoms) and the disease genotype (genotype refers to your genetic information). The investigator also wants to identify biomarkers of ALS and related diseases.

ELIGIBILITY:
Inclusion Criteria for affected individuals (primary participants) include:

* Clinical diagnosis or suspicion of ALS or a related disorder, including, but not limited to, ALS-FTD, PLS, HSP, FTD, Multisystem Proteinopathy (MSP) and PMA.
* Subject is able and willing to comply with study procedures

Exclusion Criteria for affected individuals (primary participants) include:

* Subjects with a condition or who are in a situation which, in the PI's opinion, could confound the study finding or may interfere significantly with the individual's participation and compliance with the study protocol -- including but not limited to neurological, psychological and/or medical conditions

Inclusion criteria for biological family members (secondary participants) include:

* Family member of an enrolled affected primary participant

Exclusion Criteria for biological family members (secondary participants) include:

* Subjects with a condition or who are in a situation which, in the PI's opinion, could confound the study finding or may interfere significantly with the individual's participation and compliance with the study protocol -- including but not limited to neurological, psychological and/or medical conditions

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary participants - patients that have or are suspected to have ALS or a related disease.
  Secondary participants - family members of primary participants enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Rates of change in revised ALS functional rating scale (ALSFRS-R) | 48 months
  Prepare motor outcome measures for clinical trials in sub-populations of patients with ALS or a related disorder who have identifiable genetic causes of disease
Rates of change in Slow vital capacity (SVC) | 48 months
  Prepare motor outcome measures for clinical trials in sub-populations of patients with ALS or a related disorder who have identifiable genetic causes of disease
Rates of change in Spastic paraplegia rating scale (SPRS) | 48 months
  Prepare cognitive and behavioral outcome measures for clinical trials in sub-populations of patients with ALS or a related disorder who have identifiable genetic causes of disease
Rates of change in Edinburgh Cognitive and Behavioral ALS Screen (ECAS) | 48 months
  Prepare cognitive and behavioral outcome measures for clinical trials in sub-populations of patients with ALS or a related disorder who have identifiable genetic causes of disease
ALS Health Index (ALS-HI) | 48 months
  Validate the ALS Health Index (ALS-HI), a novel patient reported outcome (PRO) measure
Serum | 48 months
  Determine the diagnostic utility of serum neurofilament concentrations
Cerebrospinal Fluid (CSF) | 48 months
  Determine the diagnostic utility of CSF neurofilament concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Michael Benatar, MD, PhD, Principal Investigator — University of Miami
Locations (4):
- United States (3):
  - University of Miami, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Pennsylvania, Philadelphia, Pennsylvania
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No